CLINICAL TRIAL: NCT01626729
Title: Facts-Up-Front Versus Traffic-Light Food Labels: A Randomized Controlled Trial
Brief Title: Facts-Up-Front Versus Traffic-Light Food Labels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, Christina Roberto, Principal Investigator, Yale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1101007870
Record Dates: First submitted 2012-06-14; First posted 2012-06-25 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Food Labeling
Keywords: Food Labeling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Traffic Light (Experimental)
  Interventions: Behavioral: Traffic Light
- Traffic Light+ (Experimental)
  Interventions: Behavioral: Traffic Light+
- Facts Up Front (Experimental)
  Interventions: Behavioral: Facts Up Front
- Facts Up Front+ (Experimental)
  Interventions: Behavioral: Facts Up Front+
- No front of package label (Placebo Comparator)
  Interventions: Behavioral: No label control group

INTERVENTIONS:
Behavioral: Traffic Light — A kilocalories (calories) per serving label and a Traffic Light symbol with High/Med/Low text indicating amounts of saturated fat, total sugars, and sodium per serving.
  Arms: Traffic Light
Behavioral: Traffic Light+ — A calories per serving label and a Traffic Light symbol with High/Med/Low text indicating amounts of saturated fat, total sugars, sodium, fiber and protein per serving.
  Arms: Traffic Light+
Behavioral: Facts Up Front — A label displaying calories, saturated fat, sodium, and total sugars per serving. Nutrient amounts were listed in grams/milligrams and % Daily Values (%DVs), which indicate whether a serving of food is high or low in a nutrient based on daily value recommendations for a 2,000 calorie diet, were included. This symbol was created based on the Facts Up Front symbol description provided by the Grocery Manufacturers Association and Food Marketing Institute, without the inclusion of nutrients to encourage.
  Arms: Facts Up Front
Behavioral: Facts Up Front+ — A label displaying calories, saturated fat, sodium, and total sugars per serving. The label also showed two (out of the possible eight) nutrients to encourage with the highest %DV. Nutrient amounts were listed in grams/milligrams and %DVs were included. This symbol was based directly on the Facts Up Front symbol description provided by the Grocery Manufacturers Association and Food Marketing Institute.
  Arms: Facts Up Front+
Behavioral: No label control group — No label control group
  Arms: No front of package label

SUMMARY:
The U.S. food and beverage industry recently released a new front-of-package nutrition labeling system called Facts Up Front that will be used on thousands of food products. The purpose of this study was to test consumer understanding of the Facts Up Front nutrition labeling system compared to the Multiple Traffic Light system (Traffic Light). Facts Up Front displays grams/milligrams and % daily value information for various nutrients; Traffic Light uses an interpretive color-coded scheme to alert consumers to low, medium or high levels of certain nutrients. Participants in an Internet-based study were randomized to one of five front-of-package label conditions: 1) No Label; 2) Traffic Light; 3) Traffic Light plus information about protein and fiber (Traffic Light+); 4) Facts Up Front; or 5) Facts Up Front plus information about "nutrients to encourage" (Facts Up Front+). Total percentage correct quiz scores were generated reflecting participants' ability to compare two foods on nutrient levels, based on their labels, and to estimate amounts of saturated fat, sugar, sodium, fiber and protein in foods. 703 adult participants recruited through an online database in May 2011 participated in this Internet-based study and data were analyzed in June 2011. The investigators hypothesized that the Traffic Light label groups would perform better than the Facts Up Front groups on all outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participants in Survey Sampling International Panels

Exclusion Criteria:

* Younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 703 (Actual)
Dates: Start 2011-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Nutrient Comparison and Nutrient Level Estimation Accuracy | Baseline
  Participants took a nutrient level comparison quiz asking them to identify which of two products presented side-by-side in the same food category were higher or lower in different nutrients. Participants also viewed 8 individual products and estimated whether the product had low, medium or high amounts of saturated fat, sugar, sodium, fiber, and protein. The primary outcomes were total percentage correct on these quizzes.
Perceptions of Health, Taste and Purchase Intent | Baseline
  Participants rated how healthy they thought each individual product was, how good it would taste and their likelihood to buy the product for themselves and their children (answered only by those who reported having children) using a 9-point Likert scale. Each set of ratings was averaged across eight products.

SECONDARY OUTCOMES:
Consumer Label Preferences | Baseline
  Composite scores were created based on several items assessing ease of label interpretation and understanding, label complexity, and degree of label confusion.

CONTACTS AND LOCATIONS:
Overall Officials: Christina A Roberto, PhD, Principal Investigator — Yale University
Locations (1):
- Survey Sampling International & Yale University, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Roberto CA, Bragg MA, Schwartz MB, Seamans MJ, Musicus A, Novak N, Brownell KD. Facts up front versus traffic light food labels: a randomized controlled trial. Am J Prev Med. 2012 Aug;43(2):134-41. doi: 10.1016/j.amepre.2012.04.022. PMID 22813677